CLINICAL TRIAL: NCT04017182
Title: Correlation Between External Jugular Venous and Superior Vena Cava Central Venous Blood Oxygen Saturation in Patient Under General Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Thanist Pravitharangul, Principal investigator, Ramathibodi Hospital
Other Study IDs: 04072019
Record Dates: First submitted 2019-07-04; First posted 2019-07-12 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Central Venous Oxygen Saturation
Keywords: central venous oxygen saturation; external jugular venous oxygen saturation; central venous catheter; external jugular vein; internal jugular vein; superior vena cava oxygen saturation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
After installation of central venous catheter in patients under general anesthesia, paired sample of superior vena cava central venous blood and right external jugular venous blood will be collected and send to central laboratory for venous blood gas analysis. Correlation between superior vena cava central venous blood and right external jugular venous blood oxygen saturation will be determined as primary outcome.

DETAILED DESCRIPTION:
All patients age between 18-65 year old who undergoing surgery under general anesthesia and superior vena cava central venous catheter installation anticipated are eligible. The tips of superior vena cava central venous catheter was confirmed by Chest x-ray. Next 1 hour after skin incision, 1 ml of venous blood sample is taken from superior vena cava central venous catheter of right external jugular vein then send to central laboratory for venous blood gas analysis. The demographic data will be recorded. Correlation between superior vena cava central venous blood and right external jugular venous blood oxygen saturation will be determined the primary outcome and partial pressure of carbon dioxide will be determined as a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Written consent obtained from patient or next of kin a day before operation date
* Patient age between 18-65 years old undergoing syrgery under general anesthesia
* Superior vena cava central venous catheter anticipated for CVP mesurement, innotropic or vasopressor administration,pulmonary artery catheter insertion route
* Anticipated right external jugular venous sampling time less than 5 minutes
* The site of blood sample collection easily access during operation

Exclusion Criteria:

* No jugular central venous catheter installation or other route selected
* Duration of paired sample collection more than 10 minutes
* Can not collected blood sample from right external jugular vein within 3 attemps
* The site of blood sample collection difficulty access during operation
* Pateint or next of kin refuse to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult surgical patients undergoing surgery under general anesthesia in institutional operating theaters with superior vena cava central venous catheter installation anticipated.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of venous oxygen saturation | 1 hour
  Correlation of venous oxygen saturation between external jugular vein and superior vena cava

SECONDARY OUTCOMES:
Correlation of venous partial pressure of carbon dioxide | 1 hour
  Correlation of venous partial pressure of carbon dioxide between external jugular vein and superior vena cava
Relationship between superior vena cava central venous and external jugular venous oxygen saturation | 1 hour
  Linear regression to determine prediction equation between superior vena cava oxygen saturation and external jugular vein oxygen saturation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Ramathibodi Hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No